CLINICAL TRIAL: NCT04027933
Title: An Examination of the Education Based on Standard Patient Simulation in Nursing Students' Approach Toward Patients With Bipolar Disorder: Randomized Controlled Research
Brief Title: Standard Patient Simulation in Nursing Students' Approach Toward Patients With Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Nesibe Gunay Molu, Director, Nursing Department, Principal Investigator and Phd student, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Nesibe GUNAY MOLU
Record Dates: First submitted 2019-07-02; First posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Educational Problems; Anxiety and Fear; Nurse-Patient Relations
Keywords: Psychiatric nursing; Simulation; Standardized patients
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Two parallel group pretest-poshest randomized control trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor does not know which group the data belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Active Comparator): Education Based on Standard Patient Simulation was given to this group
  Interventions: Behavioral: Education Based on Standard Patient Simulation
- Control (No Intervention): Control group

INTERVENTIONS:
Behavioral: Education Based on Standard Patient Simulation — In the first phase of the study, a theoretical education was provided to the students.
  In the second phase, the students in the experimental and control groups who completed their theoretical education were given data collection forms. In the third phase, after the scales were implemented, there was no intervention with the control group. There was a standard patient implementation to the experimental group. In the fourth phase of the study, after completing the simulation practice, all scales were re-applied both to the experimental and control groups. The scales were applied after the simulation training was completed and students were sent to the clinical practice after three weeks. In the fourth phase of the study, right before the students practiced their trainings and at the end of the initial rotations of the clinical practice, which turned out to be about four weeks later on average, all scales were re-applied both to the experimental and control groups.
  Arms: Experimental

SUMMARY:
The study was conducted to determine the effect of the simulation method with the participation of standardized patients towards the patients suffering from bipolar disorder to benefit the education of the psychiatry nursing students.

The Research Questions

1. Does the use of simulation training with the standardized patients have any effect on the average scores of the fear and behavioral intentions of the students as they approach patients with bipolar disorder?
2. Does the use of simulation training with the standardized patients have any effect on the average scores of the communication skills assessment scale of the students as they approach patients with bipolar disorder?
3. Does the use of simulation training with the standardized patients have any effect on the average scores of the state and trait anxiety level of the students as they approach patients with bipolar disorder?
4. Does the use of simulation training with the standardized patients have any effect on the average scores of the clinical decision making in the nursing scale of the students as they approach patients with bipolar disorder?
5. Does the use of simulation training with the standardized patients have any effect on the average scores of the self-efficacy - sufficiency scale of the students as they approach patients with bipolar disorder?

DETAILED DESCRIPTION:
The students of the Department of Nursing in the Faculty of Health Sciences at Ankara's Yıldırım Beyazıt University during the 2017-2018 academic year constitute the research universe. The research universe was randomly selected from the students who voluntarily accepted to participate in the research and met the research criteria. The Minitab software was used to calculate samples and 99% confidence interval with type 1 error 0.05 was accepted. A 0.5 score difference of the anxiety scale was accepted as a success and a sample of 76 students with 38 in the experimental and 38 in the control group was agreed upon. This calculation was based on the change in the anxiety scale score after the simulation education in Kameg et al.'s 2014 study. The power analysis at the end of the study indicated that the scale's average scores ranged between 0.56-0.98. Foreign national students were not included in the study in order to generate a common language. 83 students who will be trainees in the psychiatric clinics and community mental health centers (CMHC) were included in the study and constituted the experimental and control groups. Female and male students were ranked from the highest to the lowest by their academic success scores, and random numbers were assigned in excel to randomly divide these ranked students among the groups. This randomization procedure was done in class. Numbers greater than 0.5 were assigned to the experimental group and numbers lower than 0.5 were assigned to the control group.

Before the study began, two students whose clinical practice locations had changed and two students who were absent in the theoretical class were excluded from the study, and 79 students were divided into two groups as 40 students for the experimental and 39 students for the control group. In the experimental group, 2 students who were absent in the simulation practice and one student who did not properly fill out the data collection form were excluded from the study. In the control group, two students who did not want to fill out the data collection form were also excluded from the study. The study was completed with 37 students from experimental group and 37 from the control group - 74 individuals in total.

Data Evaluation The research data was evaluated in SPSS 22.0 statistical software as appropriate to the quality of the data and research. Normality analysis was conducted by Kolmogorov Smirnov, Shapiro-Wilk, skewness and kurtosis values.

To evaluate the impact size of the education program, variance analysis was used in the repeating assessment. In this study, the impact size of the education was found 1.45≤, and evaluated as very high levels.

ELIGIBILITY:
Inclusion Criteria:

• Volunteer Students

Exclusion Criteria:

• Foreign National Students

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2017-11-23 (Actual); Study Completion 2017-11-23 (Actual)

PRIMARY OUTCOMES:
Fear and Behavior Intent Scale | Change from fear and behavioral intentions of the students at 2 months.
  The scale, developed by Wolf (1996) measures fear and behavioral attitudes toward mentally disordered patients. The scale was adapted into Turkish by Günay Molu and Özkan after the required permission was taken from the e-mail address on the original article (Günay Molu and Özkan 2018). It is a 5-Likert type scale including ten items, and each item is graded between 1-5. An change in the total score of the scale means an change in negative attitudes towards the mentally disordered patient. Cronbach's alpha was 0.784.
The Communication Skills Assessment Scale | Change from communication skills assessment scale of the students at 2 months.
  The 5-Likert type scale developed by Korkut (1996) is scored from "always" to "never". The scale consists of 25 items in total, and the maximum possible score is 100 while zero is the minimum. Higher scores indicate better communication skills. The reliability coefficient is .76 and the alpha internal consistency coefficient is .80.
State and Trait Anxiety Level | Change from the state and trait anxiety level of the students at 2 months.
  The scale developed by Spielberger in 1970 is a self-assessment questionnaire which is used to define state and trait anxiety levels. It was adapted into Turkish by Öner and Le Compte in 1985. It is a 4-Likert type scale. The scores of both scales range from 20 to 80 in total (Oner, 1992). It is reported that the Alpha's coefficient ranges between .83 and .87, while the test re-test reliability ranges between .71 and .86, and the item reliability ranges between .34 and .72.
Self-Efficacy - Sufficiency Scale | Change from the self-efficacy - sufficiency scale of the students at 2 months.
  The scale developed by Sherer et al. (1982) and adapted into Turkish by Gözüm and Aksayan (1999) was developed to assess behavior and behavioral changes. It is a 23 item 5-Likert type self-assessment scale. Its score ranges between 23 and 115. Higher scores mean that the individual has higher SES perception (Gözüm and Aksayan, 1999). The reliability and validity of the Turkish version was done for the same sample, and the Cronbach's alpha internal consistency coefficient was found to be .81, and the test re-test reliability was .92.
Clinical Decision Making in The Nursing Scale | Change from the clinical decision making in the nursing scale of the students at 2 months.
  The scale developed by Jenkins (1983) defines the clinical decision making perceptions of nursing students. The original scale consists of 40 items and four sub-scales. Each sub-scale consists of 10 items. Total score ranges between 40 and 200, and each subscale ranges between 10 and 50 with no cut-off point. Total Cronbach's alpha reliability coefficient is 0.78.

CONTACTS AND LOCATIONS:
Overall Officials: Birgül Özkan, Assoc. Prof, Study Director — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yıldırım Beyazıt Universty, Faculty Of Health Sciences, Department Nursing, Mental health and Nursing, Ankara, Turkey (Türkiye)